CLINICAL TRIAL: NCT02260245
Title: Stepping Up for Safety: Improving Teamwork at the Planned Parenthood Affiliates Through the TeamSTEPPS Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Affiliates Risk Management Services, Inc. (Industry)
Responsible Party: Principal Investigator, Maureen Paul, Division Director of Family Planning, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014P000045
Record Dates: First submitted 2014-09-25; First posted 2014-10-09 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Improving Team Work at the Planned Parenthood Affiliates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Team training (Other): All participating affiliates will undergo team training using the TeamSTEPPS model
  Interventions: Behavioral: Team training using the TeamSTEPPS model

INTERVENTIONS:
Behavioral: Team training using the TeamSTEPPS model — Two or three master trainers from each affiliate will be undergo train-the-trainer training to bring back to their affiliate.

SUMMARY:
TeamSTEPPS (Team Strategies and Tools to Enhance Performance and Patient Safety) is an evidence-based teamwork system designed to improve communication and teamwork skills among health professionals. The program was developed by the Agency for Healthcare Research and Quality (AHRQ) and the Department of Defense's Patient Safety Program as the national standard for team training in health care.

The purpose of this study is to evaluate the effect of the TeamSTEPPS program on the team knowledge, skills and attitudes and patient safety at Planned Parenthood affiliates nationwide.

The investigators hypothesize that implementation of the TeamSTEPPS program will be associated with improved team knowledge, skills, and attitudes; clinical outcomes; and process outcomes.

Aims:

1. To assess the effect of the TeamSTEPPS training program on team communication and effective team work
2. To assess the effect of the TeamSTEPPS training program on process outcomes
3. To assess the effect of the TeamSTEPPS training program on clinical outcomes

DETAILED DESCRIPTION:
In 1999, the healthcare community received a wake-up call when the Institute of Medicine's landmark report, To Err Is Human, [IOM, 1999] revealed that up to 98,000 Americans die each year from medical errors, with several more thousand injured. Most medical errors result from systems deficiencies, and they include such events as missed or delayed diagnoses and medication errors. The morbidity, mortality, and associated costs that result from medical errors can have far-reaching consequences, not only for patients and their families, but also for caregivers, health care organizations, and the community at large.

Publication of the IOM report heralded a seismic shift in the culture and delivery of health care as medical facilities sought to identify and redesign vulnerable systems to make them safer. Most efforts to date have concentrated on hospital-based systems, however, and a tremendous need exists to adapt "lessons learned" and patient safety strategies and tools to ambulatory-care facilities [Sclafani 2012]. Toward that end, Affiliates Risk Management Services, Inc. (ARMS), the risk management foundation for Planned Parenthood of America (PPFA), is partnering with Beth Israel Deaconess Medical Center/Harvard Medical School (BIDMC/HMS) and the Agency for Healthcare Research and Quality (AHRQ) to bring team training to PPFA's large clinical network. This network is comprised of 74 affiliates operating ambulatory health centers throughout the United States that provide reproductive health services to approximately 3 million women and men annually.

Implementation of a medical teamwork system has been associated with reduced medical errors, improved clinical and process outcomes, and medical and liability cost savings [Colla 2005; Mann 2006; Pratt 2007; Neilsen 2007, Neily 2010; Gillespie 2010; Weaver 2010; Moffatt 2012; Gluck 2012; Sawyer 2013]. For example, in a recent large study involving more than 100,000 surgical procedures in 100 Veterans Administration hospitals, patients whose surgical staff had undergone team training experienced a 50% greater decline in surgical mortality than those whose staff had not been team-trained [Neily 2010]. In a seminal study at BIDMC/HMS, implementation of a team training initiative among labor and delivery staff resulted in a 50% decrease both in the incidence of adverse obstetrical outcomes and the number of high severity malpractice claims, representing a savings of several million dollars [Mann 2006, Pratt 2007]. Team training results in higher quality, safer care by producing high performing teams, clarifying roles and responsibilities, improving information sharing, and eliminating barriers to quality and safety. Moreover, team training has the potential to help shift the organizational culture of health care institutions from hierarchical models to ones that foster team learning, collaboration, transparency, and open communication.

The move toward greater safety in health care is not only the "right thing to do" for patients, but it has become a national imperative. Nearly half of The Joint Commission's standards for accreditation of health care facilities directly relate to patient safety [The Joint Commission, online 2013], and effective communication and team work are key components of the American Congress of Obstetricians and Gynecologists' [ACOG] recently-launched voluntary accreditation program for medical office settings [Sclafani et al. 2012]. Indeed, the ability to thrive in the new environment of health care reform demands delivery of care that is safe, high-quality, efficient, and cost-effective, all characteristics affected by team training. The time has come to bring the benefits of team training to the Planned Parenthood network and the myriad patients who turn to Planned Parenthood as their trusted health care provider.

This is a prospective cohort study to evaluate the effect of the TeamSTEPPS program on team knowledge, skills and attitudes, process outcomes, and clinical outcomes in Planned Parenthood affiliates in the United States.

Study Population: Planned Parenthood affiliate employees and clients will serve as the study population for this study. Some endpoints, such as attitudes about team work, will rely on client and employee surveys pre- and post-intervention. Process outcomes such as frequency of team briefs will rely on affiliate documentation of the frequency of these events pre- and post-intervention. Clinical outcomes, such as adverse events, will utilize the secure online de-identified reporting system, ARMS Risk Management Information System (AIMS).

Intervention: During a two-year period, ARMS/BIDMC plans to offer TeamSTEPPS master training for key staff from 16 Planned Parenthood affiliates and to assist these master trainers as they implement targeted improvements through team training at the affiliate level. TeamSTEPPS, an evidence-based teamwork system designed to improve communication and teamwork skills among health professionals, was developed by AHRQ and the Department of Defense's Patient Safety Program as the national standard for team training in health care [AHRQ on line; Sheppard et al. 2013]. Faculty members from AHRQ's TeamSTEPPS national training center at the University of Washington have agreed to provide a dedicated master training course for Planned Parenthood affiliates. ARMS will work with the faculty to adapt the TeamSTEPPS curriculum to the Planned Parenthood clinical context.

Procedures:

The training and implementation cycle includes the following main components that are occurring independent of the evaluation:

1. Developing a Teamwork Improvement Action Plan Using a guide developed by AHRQ, ARMS staff and BIDMC/HMS faculty will work with each participating affiliate to develop a Teamwork Improvement Action Plan prior to the master training program. The purpose is to help each affiliate prepare for team training by identifying an appropriate training team and determining two to three key targets for improvement through team training, how the intervention will be implemented, and how to measure success.
2. TeamSTEPPS Master Training Each of the selected affiliates will send a 2-4 person team to a 2-day TeamSTEPPS "train the trainer" program in June 2014. The teams will be multidisciplinary (for example, quality leader, physician, nurse manager) and consist of leaders who are well-positioned by their roles to offer team training to frontline surgical abortion staff at their affiliates.

   The training curriculum teaches practical tools and strategies, such as briefs, huddles, debriefs, time outs, and SBAR (situation - background - assessment - recommendation) communication skills that when practiced regularly, cultivate the core team skills necessary for effective team work.
3. TeamSTEPPS Implementation at the Clinic Level Following the master training, the TeamSTEPPS master trainers will implement their Action Plans at their affiliates.
4. Continued Training and Sustainability ARMS staff will advise and support the new master trainers as they reinforce the principles and skills of TeamSTEPPS on an ongoing basis. In addition, the trainers will be encouraged to participate in AHRQ's TeamSTEPPS user support network, which includes web conferences and an online discussion forum, as well as AHRQ's annual TeamSTEPPS national conference.

ELIGIBILITY:
Inclusion Criteria:

* Planned Parenthood employee
* Planned Parenthood client

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Change in team attitudes and perceptions | Pre-intervention, six months post-intervention, and every 12 months thereafter
  Surveys will be completed by staff at each affiliate; additional surveys will be completed anonymously by patients regarding their perceptions of teamwork among the affiliate staff members involved in their care. These measures will be used to create a composite measure, and change from baseline to each of the study time-points will be assessed.
Change in process outcomes and behavioral change | Pre-intervention, six months post-intervention, and every 12 months thereafter
  A designated staff member at each affiliate will complete a questionnaire regarding site practices such as the use of time-outs and the occurrence of briefs and debriefs. These outcomes will be combined as a composite measure, and change from baseline to each of the study time-points will be assessed.
Change in clinical outcomes | Pre-intervention, six months post-intervention, and every 12 months thereafter
  Adverse outcomes are collected by AIMS and will be reported in a de-identified report to the research team. All adverse outcomes will be combined to create a composite measure, and change from baseline to each of the study time-points will be assessed.
Change in patient cycle times | Six-month period before intervention and for six months after a six-month washout period after intervention
  Organizations track the time that patients spend in the clinic such that changes in patient cycle time (intake to exit) can be measured

CONTACTS AND LOCATIONS:
Overall Officials: Maureen E Paul, MD, Principal Investigator — Beth Israel Deaconess Medical Center

REFERENCES:
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America; Kohn LT, Corrigan JM, Donaldson MS, editors. To Err is Human: Building a Safer Health System. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK225182/ PMID 25077248
- [Background] Sclafani J, Levy B, Lawrence H, Saraco M, Cain JM. Building a better safety net: taking the safety agenda to office-based women's health. Obstet Gynecol. 2012 Aug;120(2 Pt 1):355-9. doi: 10.1097/AOG.0b013e318260957c. PMID 22668586
- [Background] Colla JB, Bracken AC, Kinney LM, Weeks WB. Measuring patient safety climate: a review of surveys. Qual Saf Health Care. 2005 Oct;14(5):364-6. doi: 10.1136/qshc.2005.014217. PMID 16195571
- [Background] Pratt SD, Mann S, Salisbury M, Greenberg P, Marcus R, Stabile B, McNamee P, Nielsen P, Sachs BP. John M. Eisenberg Patient Safety and Quality Awards. Impact of CRM-based training on obstetric outcomes and clinicians' patient safety attitudes. Jt Comm J Qual Patient Saf. 2007 Dec;33(12):720-5. doi: 10.1016/s1553-7250(07)33086-9. No abstract available. PMID 18200896
- [Background] Nielsen PE, Goldman MB, Mann S, Shapiro DE, Marcus RG, Pratt SD, Greenberg P, McNamee P, Salisbury M, Birnbach DJ, Gluck PA, Pearlman MD, King H, Tornberg DN, Sachs BP. Effects of teamwork training on adverse outcomes and process of care in labor and delivery: a randomized controlled trial. Obstet Gynecol. 2007 Jan;109(1):48-55. doi: 10.1097/01.AOG.0000250900.53126.c2. PMID 17197587
- [Background] Neily J, Mills PD, Young-Xu Y, Carney BT, West P, Berger DH, Mazzia LM, Paull DE, Bagian JP. Association between implementation of a medical team training program and surgical mortality. JAMA. 2010 Oct 20;304(15):1693-700. doi: 10.1001/jama.2010.1506. PMID 20959579
- [Background] Gillespie BM, Chaboyer W, Murray P. Enhancing communication in surgery through team training interventions: a systematic literature review. AORN J. 2010 Dec;92(6):642-57. doi: 10.1016/j.aorn.2010.02.015. PMID 21130202
- [Background] Moffatt-Bruce SD, Funai EF, Nash M, Gabbe SG. Patient safety strategies: are we on the same team? Obstet Gynecol. 2012 Oct;120(4):743-5. doi: 10.1097/AOG.0b013e31826af730. No abstract available. PMID 22996089
- [Background] Gluck PA. Patient safety: some progress and many challenges. Obstet Gynecol. 2012 Nov;120(5):1149-59. doi: 10.1097/aog.0b013e31826feaa0. PMID 23090534
- [Background] Sawyer T, Laubach VA, Hudak J, Yamamura K, Pocrnich A. Improvements in teamwork during neonatal resuscitation after interprofessional TeamSTEPPS training. Neonatal Netw. 2013 Jan-Feb;32(1):26-33. doi: 10.1891/0730-0832.32.1.26. PMID 23318204
- [Background] Weaver SJ, Rosen MA, DiazGranados D, Lazzara EH, Lyons R, Salas E, Knych SA, McKeever M, Adler L, Barker M, King HB. Does teamwork improve performance in the operating room? A multilevel evaluation. Jt Comm J Qual Patient Saf. 2010 Mar;36(3):133-42. doi: 10.1016/s1553-7250(10)36022-3. PMID 20235415
- [Background] Sheppard F, Williams M, Klein VR. TeamSTEPPS and patient safety in healthcare. J Healthc Risk Manag. 2013;32(3):5-10. doi: 10.1002/jhrm.21099. PMID 23335296
- [Background] Baker DP, Amodeo AM, Krokos KJ, Slonim A, Herrera H. Assessing teamwork attitudes in healthcare: development of the TeamSTEPPS teamwork attitudes questionnaire. Qual Saf Health Care. 2010 Dec;19(6):e49. doi: 10.1136/qshc.2009.036129. Epub 2010 Aug 10. PMID 20702444
- [Background] Castner J. Validity and reliability of the Brief TeamSTEPPS Teamwork Perceptions Questionnaire. J Nurs Meas. 2012;20(3):186-98. doi: 10.1891/1061-3749.20.3.186. PMID 23362556
- [Background] Mann S, Marcus R, Sachs B. Lessons from the cockpit: How team training can reduce errors on L&D. Contemp OB/GYN, January 2006, p. 1-7.
- [Background] Agency for Healthcare Research and Quality (AHRQ). TeamSTEPPS: National Implementation. Rockville MD: AHRQ. Available at teamstepps.ahrq.gov. Accessed February 1, 2013.